CLINICAL TRIAL: NCT03458845
Title: Prevalence of Sarcopenia and Undernutrition in Patients With Cirrhosis and Abdominal Hernia
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Alberto Meyer, MD PhD FACS, Principal Investigator, University of Sao Paulo
Other Study IDs: 81063817.0.0000.0068
Record Dates: First submitted 2018-02-26; First posted 2018-03-08 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Cirrhosis; Sarcopenia; Malnutrition; Hernia, Abdominal
Keywords: Cirrhosis; Sarcopenia; Malnutrition; Inguinal hernia; Umbilical hernia; Undernutrition
MeSH Terms: conditions — Fibrosis; Sarcopenia; Malnutrition; Hernia, Abdominal; Hernia, Inguinal; Hernia, Umbilical | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: This group consists of cirrhotic patients with any abdominal hernia
  Interventions: Diagnostic Test: Computed Tomography Scan
- Group 2: This group consists of cirrhotic patients without any hernias
  Interventions: Diagnostic Test: Computed Tomography Scan

INTERVENTIONS:
Diagnostic Test: Computed Tomography Scan — The results of the CT scan and the hand-grip test will be used for diagnosis of sarcopenia. The Royal Free Hospital-Global Assessment (RFH-GA) results will classify the nutritional status of the patient.
  Other Names: Hand-grip test (dynamometer); Royal Free Hospital-Global Assessment

SUMMARY:
The study evaluates whether sarcopenia influences the prevalence of abdominal hernias in patients with cirrhosis.

DETAILED DESCRIPTION:
Sarcopenia is a common condition in patients with cirrhosis, with a prevalence of around 50%. It is unknown if the presence of sarcopenia may influence the prevalence of abdominal hernias in this group of patients. Clinical, nutritional and radiological evaluation will be performed in two groups of cirrhotic patients to evaluate this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Previous diagnosis of cirrhosis

Exclusion Criteria:

* Acutely decompensated cirrhosis
* Other chronic diseases in advanced stage (e.g. cardiac failure, chronic obstructive pulmonary disease, cancer)
* Cognitive impairment, delirium, non-controlled psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary care adult patients with cirrhosis, with and without abdominal hernias.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of Sarcopenia | Through study completion (an average of 1 year)
  Prevalence of Sarcopenia in patients with cirrhosis
Influence of Sarcopenia in Prevalence of Abdominal Hernias in Patients with Cirrhosis | Through study completion (an average of 1 year)
  Influence of Sarcopenia in Prevalence of Abdominal Hernias in Patients with Cirrhosis

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Meyer, PhD, Principal Investigator — Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Montano-Loza AJ. Clinical relevance of sarcopenia in patients with cirrhosis. World J Gastroenterol. 2014 Jul 7;20(25):8061-71. doi: 10.3748/wjg.v20.i25.8061. PMID 25009378
- [Background] Kalafateli M, Konstantakis C, Thomopoulos K, Triantos C. Impact of muscle wasting on survival in patients with liver cirrhosis. World J Gastroenterol. 2015 Jun 28;21(24):7357-61. doi: 10.3748/wjg.v21.i24.7357. PMID 26139982
- [Background] Morgan MY, Madden AM, Soulsby CT, Morris RW. Derivation and validation of a new global method for assessing nutritional status in patients with cirrhosis. Hepatology. 2006 Oct;44(4):823-35. doi: 10.1002/hep.21358. PMID 17006918
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703